CLINICAL TRIAL: NCT06138444
Title: A Randomized Controlled Clinical Trial of Cordyceps Militaris Beverage on the Immune Response
Brief Title: Effect of Cordyceps Militaris Beverage on the Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Phayao (Other)
Collaborators: National Innovation Agency (NIA) (Unknown)
Responsible Party: Principal Investigator, Atcharaporn Ontawong, Assistant Professor Dr., University of Phayao
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UP-HEC 1.3/026/65
Record Dates: First submitted 2023-10-17; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Cordyceps militaris; Healthy subjects; NK cell; Cytokine; Immunomodulation
MeSH Terms: interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Intervention Model Description: Male or female received a single oral dose of functional beverages from submerged fermentation of Cordyceps militaris (FCM) or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Male received functional beverages (Experimental): Male received single oral dose of functional beverages from submerged fermentation of Cordyceps militaris (FCM)
  Interventions: Dietary Supplement: Functional beverages from the submerged fermentation of Cordyceps militaris
- Male received placebo (Placebo Comparator): Male received placebo
  Interventions: Other: Fruit juice
- Female received functional beverages (Experimental): Female received single oral dose of functional beverages from submerged fermentation of Cordyceps militaris (FCM)
  Interventions: Dietary Supplement: Functional beverages from the submerged fermentation of Cordyceps militaris
- Female received placebo (Placebo Comparator): Female received placebo
  Interventions: Other: Fruit juice

INTERVENTIONS:
Dietary Supplement: Functional beverages from the submerged fermentation of Cordyceps militaris — The Cordyceps militaris submerged fermentation in fruit juice.
  Other Names: FCM
  Arms: Female received functional beverages; Male received functional beverages
Other: Fruit juice — Fruit juice is used as a placebo.
  Other Names: Placebo
  Arms: Female received placebo; Male received placebo

SUMMARY:
This study developed functional beverages from the submerged fermentation of Cordyceps militaris (FCM) and aimed to investigate the potential of FCM in male and female healthy volunteers in Phayao province, Thailand. To provide essential information for the development of healthy drink products.

DETAILED DESCRIPTION:
Healthy Thai males and females aged 25-60 were recruited at the School of Medical Sciences, University of Phayao, in 2022. Written informed consent was obtained from all research participants. A total of 40 participants were randomly assigned to one of the study groups (10 subjects each).

Inclusion Criteria :

1. Male and female adult participants aged 25-60 during the screening test.
2. No history of hypersensitivity or idiosyncratic reactions to drugs or herbal products.
3. Willing to participate in the project throughout the research program.

Exclusion Criteria :

1. Participants diagnosed with immune-mediated disease, nervous system disorders, cardiovascular disease, or liver or kidney disease.
2. Participants diagnosed with chronic health problems such as hypertension, diabetes, or renal failure, etc.
3. A body mass index (BMI) greater than 29.9 or less than 18 kg/m2.
4. Participants who were pregnant or lactating or intended to become pregnant during the trial period.
5. Participants who, within two weeks, ingested a drug or functional food that may affect the immunomodulatory effect of the test product.
6. Participants who had an alanine transaminase (ALT) or aspartate transaminase (AST) plasma level more than three times the guideline of the organization.

Laboratory research has been conducted to confirm the eligibility of research participants, including hematology, serum biochemistry, blood coagulation, and urinalysis. The participants who met the inclusion requirements were randomized into experimental groups. Twenty random numbers were generated using Statistical Package for the Social Sciences (SPSS) 26.0. Digits 1st-10th of each gender were numbered as the FCM group, and the remaining digits, 11th-20th of each gender, were numbered as the placebo group. All researchers, participants, and related medical staff were blinded to the intervention assignments throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult participants aged 25-60 during the screening test.
* No history of hypersensitivity or idiosyncratic reactions to drugs or herbal products.
* Willing to participate in the project throughout the research program.

Exclusion Criteria:

* Participants diagnosed with immune-mediated disease, nervous system disorders, cardiovascular disease, or liver or kidney disease.
* Participants diagnosed with chronic health problems such as hypertension, diabetes, or renal failure, etc.
* A body mass index (BMI) greater than 29.9 or less than 18 kg/m2.
* Participants who were pregnant or lactating or intended to become pregnant during the trial period.
* Participants who, within two weeks, ingested a drug or functional food that may affect the immunomodulatory effect of the test product
* Participants who had an alanine transaminase (ALT) or aspartate transaminase (AST) plasma level more than three times the guideline of the organization.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change from the baseline on physical examination (Height) | At 0, 4 and 8 weeks after end of the intervention
  The first visit was conducted within one week after screening. Every 15 days after taking the test substance, the subjects were examined for height (Centimeter).
Change from the baseline on the physical examination (Weight) | At 0, 4 and 8 weeks after end of the intervention
  The first visit was conducted within one week after screening. Every 15 days after taking the test substance, the subjects were examined for weight (Kilogram).
Change from the baseline on the physical examination (Blood pressure) | At 0, 4 and 8 weeks after end of the intervention
  The first visit was conducted within one week after screening. Every 15 days after taking the test substance, the subjects were examined for blood pressure using an automatic blood pressure monitor (mmHg).
Change from the baseline on the physical examination (oxygen saturation) | At 0, 4 and 8 weeks after end of the intervention
  The first visit was conducted within one week after screening. Every 15 days after taking the test substance, the subjects were examined for oxygen saturation using a fingertip pulse oximeter (%).
Change from the baseline on the physical examination (adverse reactions) | At 0, 4 and 8 weeks after end of the intervention
  The first visit was conducted within one week after screening. Every 15 days after taking the test substance, the subjects were examined for adverse reactions (Questionnaire).
Change from the baseline on the immune response (NK cells) | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection. This experiment examined the changes in natural killer cells (NK cells), measurement by using flow cytometry-based assays.
Change from the baseline on the cluster of differentiation (CD) antigens | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection.
  This experiment examined the changes in cluster of differentiation (CD) antigens
  1. Cluster of differentiation 3 (CD3)
  2. Cluster of differentiation 4 (CD4)
  3. Cluster of differentiation 8 (CD8)
  4. B-lymphocyte antigen CD19 (CD19)
  Measurement by using flow cytometry-based assays.
Change from the baseline on the immunoglobulins | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection.
  This experiment examined the changes in immunoglobulins
  1. Immunoglobulin A (IgA)
  2. Immunoglobulin G (IgG)
  3. Immunoglobulin M (IgM)
  Measurement by using flow cytometry-based assays.
Change from the baseline on the inflammatory cytokines | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection.
  This experiment examined the changes in inflammatory markers
  1. Tumor necrosis factor alpha (TNF-α)
  2. Interleukin 1 beta (IL-1β)
  3. Interleukin 6 (IL-6)
  Measurement by using ELISA assay.
Change from the baseline on the safety parameters (Complete blood count (CBC)) | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection. This experiment examined the changes in complete blood count (CBC), measurement by using colorimetric assays.
Change from the baseline on the safety parameters (Fasting blood glucose) | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection. This experiment examined the changes in fasting blood glucose, measurement by using colorimetric assays.
Change from the baseline on the safety parameters (Plasma lipids) | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection.
  This experiment examined the changes in safety parameters
  1. Triglyceride
  2. Total cholesterol
  Measurement by using colorimetric assays.
Change from the baseline on the safety parameters (Renal function) | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection.
  This experiment examined the changes in safety parameters
  1. Creatinine
  2. Total protein
  Measurement by using colorimetric assays.
Change from the baseline on the safety parameters (Liver function) | At 0, 4 and 8 weeks after end of the intervention
  Blood samples (10 ml for each time point) were collected at 0, 30, and 60 days. The fasting blood samples were collected into plain and ethylenediamine tetraacetic acid (EDTA) tubes and delivered to the laboratory within 2 hours of collection.
  This experiment examined the changes in safety parameters
  1. Aspartate aminotransferase (AST)
  2. Alanine aminotransferase (ALT)
  Measurement by using colorimetric assays.

CONTACTS AND LOCATIONS:
Overall Officials: Atcharaporn Ontawong, Ph.D., Principal Investigator — University of Phayao
Locations (1):
- University Of Phayao, Nai Muang, Changwat Phayao, Thailand

IPD SHARING:
Plan to Share IPD: No
Prohibited from laws (contracts)